CLINICAL TRIAL: NCT06074393
Title: Caregiving in Advanced Parkinsonian Disease: A Tailored Support Group
Brief Title: Caregiving in Advanced PD: A Tailored Support Group
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Veronica Bruno, Assistant Professor. Department of Clinical Neurosciences, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB23-0949
Record Dates: First submitted 2023-09-28; First posted 2023-10-10 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: Support group; Care partners
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Intervention Model Description: The clinical trial is a prospective study analysing the effect of a tailored support group on care partner burden, coping strategies, and quality of life in care partners of patients with advanced Parkinsonian syndromes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Care partners of patients with advanced Parkinsonian Syndromes (Experimental): Care partners of patients with advanced Parkinsonian Syndromes will participate in a tailored support group
  Interventions: Behavioral: Tailored Support Group

INTERVENTIONS:
Behavioral: Tailored Support Group — Participants engage in a secure, confidential environment, sharing caregiving insights and knowledge. Expert-led sessions, lasting 90 minutes, occur biweekly for 16 weeks, held via Zoom and at the University of Calgary's Cumming School of Medicine. These sessions take place twice annually, emphasizing the structured nature of the support group. Weekly themes include self-care, adaptation, coping skills, emotions, anticipatory grief, forgiveness, mindfulness, boundaries, and closure. Care partners actively participate by sharing experiences and asking questions in each session.
  Other Names: Support Group

SUMMARY:
The goal of this study is to understand how support groups can help people who care for individuals with Parkinson's Disease and Related Disorders (PDRD). The investigators want to find answers to these questions:

* How do these support groups make caregivers feel?
* Do these support groups help caregivers cope better and improve their quality of life?

Participants in this study will join support groups where they can talk to other caregivers and learn from experts. These groups will meet every two weeks for four months, and there will be sessions on different topics like self-care, coping skills, and mindfulness. Caregivers will share their experiences and ask questions in these sessions.

Information will be collected before and after the support group meetings using surveys. These surveys will help understand how the support groups affect caregivers. Things like caregiver burden, coping strategies, and overall well-being will be measured.

The main goal is to reduce the burden on caregivers of people with PDRD and improve their quality of life. It is believed that these support groups can make a positive difference, and this study will help understand how they work.

DETAILED DESCRIPTION:
Background & Rationale:

Neurodegenerative diseases are projected to surpass cancer as the leading cause of death by 2030. Parkinson's disease prevalence in Canada was 170/100,000 in 2013/2014, and with an aging population, the number of Canadians over 40 with the disease will rise by 65% by 2030. Advanced stages of Parkinson's Disease and Related Disorders (PDRD) result in motor disability and complex non-motor symptoms, increasing demand for healthcare services. Care partners face challenges such as anxiety, managing treatments, and uncertainty, leading to negative lifestyle changes and reduced mental health.

Care partners of PDRD must manage stressors that impact their health and well-being. Existing support groups mainly focus on disease management, and neglecting care partner challenges. These pilot support groups provide an avenue for emotional and informational support, addressing care partner burdens. Structured meetings offer practical tools, solutions, and guest speakers, enhancing support group content.

Research Question & Objectives

The study aims to establish and assess support groups tailored to PDRD care partners' needs with two main objectives:

Creating a supportive environment through structured meetings. Evaluating support group effectiveness in enhancing coping, reducing burden, and improving quality of life.

Methods:

Study Design:

The study is structured around the establishment of a supportive community for individuals caring for PDRD. The primary objective is to foster connections among caregivers, enabling them to exchange personal experiences and derive shared comfort from others who comprehend the challenges associated with these conditions.

Participants engage in a secure and confidential environment, sharing narratives and insights that contribute to their collective knowledge of effective caregiving. Moreover, the support group incorporates dedicated sessions led by healthcare experts encompassing various disciplines, including physicians, nurses, psychologists, social workers, and spiritual advisors. These specialized sessions, each lasting 90 minutes, occur biweekly over a 16-week period. Hosted at the University of Calgary's Cumming School of Medicine in a hybrid structure by using Zoom as a method of assistance, these sessions occur twice annually, accentuating the recurrent and structured nature of the support group.

In each week various themes will be addressed, such as:

Self-care and Personal Health Adaptation to changes in the living situation, changing roles and navigating the system Coping skills and Resilience Emotions (embracing vulnerability, emotional identification, factual validation, counteraction, problem resolution).

Anticipatory grief Forgiveness and interconnectedness Mindfulness Establishing boundaries, attaining tranquility, and achieving closure In every session of the support group, care partners are encouraged to participate by sharing their experiences, as well as asking pertinent questions.

Data Collection:

The study employs pre- and post-participation questionnaires and measurement instruments to assess support group efficacy comprehensively using Qualtrics as a data collection tool for the surveys.

Instruments include:

Short Zarit Burden Interview (ZBI-12) to quantify caregiving impact. Brief-COPE to assess coping mechanisms. Adult Carer Quality of Life Questionnaire (AC-QoL) to measure overall well-being.

Satisfaction Survey to gather participant feedback and knowledge acquisition.

Outcomes:

Primary Outcomes:

Care Partner Burden: Assessed using ZBI-12. Coping Strategies: Evaluated with Brief-COPE scale. Quality of Life: Scrutinized using AC-QoL scale.

Secondary Outcomes:

Satisfaction with Participation: Caregiver Support Group Satisfaction Survey

The study addresses the increasing burden on care partners of individuals with PDRD. It establishes and evaluates support groups tailored to their needs to enhance coping, reduce burden, and improve quality of life. The study utilizes structured meetings, measurement instruments, and comprehensive assessments to shed light on the effects of the support groups on care partners' well-being.

ELIGIBILITY:
Inclusion Criteria:

* Care partners of individuals with a confirmed diagnosis of Parkinsonian Syndrome.
* Participants in the Calgary Movement Disorders Advanced Care pilot program (REB22-0545)

Exclusion Criteria:

* Care partners with significant cognitive impairments that hinder participation with MoCA<10 points.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-19 (Estimated); Primary Completion 2024-10-19 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Care Partner Burden: Assessed using ZBI-12. | Enrollment and at the end of the Support Group. 1 and 16 weeks.
  ZBI-12 is validated as a screening tool for advanced illness. The ZBI-12 is rated on a 12 items scale, with the severity of burden using a range of responses from 0 to 4 points per item and a total score range of 0 to 48. Scoring 0-10 is considered as a no to mild burden; 10-20, a mild to moderate burden and >20, a high burden. It measures changes in physical, emotional, social, and financial problems that can be experienced by family caregivers.
Changes in Coping Strategies: Evaluated with Brief-COPE scale. | Enrollment and at the end of the Support Group. 1 and 16 weeks.
  The Brief COPE (Coping Orientation to Problems Experienced) scale, composed of 28 items, each rated on a 4-point scale where 3 represents the highest score, exhibits a minimum value of 0 and a maximum value of 84. When interpreting Brief COPE scores, higher values are indicative of a potentially enhanced capacity to navigate stress and handle challenging situations. These elevated scores reflect a greater propensity to employ diverse coping strategies when confronted with difficulties.
Changes in Quality of Life: Scrutinized using AC-QoL scale. | Enrollment and at the end of the Support Group. 1 and 16 weeks.
  The Adult Carer Quality of Life (AC-QoL) Scale encompasses both an overall scale and eight subscales. The overall scale yields scores ranging from 0 to 120, with higher scores signifying an enhanced quality of life for caregivers. Additionally, each of the eight subscales offers scores within a potential range of 0 to 15. Higher scores on these subscales indicate an improved quality of life for caregivers in specific domains pertaining to their caregiving responsibilities. This structured assessment provides valuable insights into the well-being of caregivers across multiple dimensions of their lives.

SECONDARY OUTCOMES:
Satisfaction with Participation: Caregiver Support Group Satisfaction Survey | Byweekly for 16 weeks
  The Caregiver Support Group Satisfaction Survey is composed of a combination of six multiple-choice questions and three open-ended questions. Each of the six multiple-choice questions is evaluated on a scale ranging from 1 to 5, with 1 signifying the lowest level of satisfaction and 5 indicating the highest level of satisfaction. Consequently, the survey's maximum achievable score is 30, while the minimum score is 5. A higher score on this survey reflects an increased level of satisfaction with the support group, providing valuable feedback on the quality of support and services offered to caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Bruno, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- Health Science Centre, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No